CLINICAL TRIAL: NCT00495677
Title: A Randomised, Double-Blind, Placebo-Controlled, Multicentre Study In Asymptomatic Hiv-Infected Patients To Investigate The Pharmacodynamics, Pharmacokinetics, Safety And Toleration Of PF-00232798
Brief Title: A Phase 2 Study Of PF-00232798 In HIV Positive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A7691009
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Results first posted 2013-10-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-08

CONDITIONS: HIV
Keywords: Treatment Experienced; Treatment Naive
MeSH Terms: interventions — PF 232798

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- PF-00232798 40 mg (Active Comparator)
  Interventions: Drug: PF-00232798
- PF-00232798 300 mg (Active Comparator)
  Interventions: Drug: PF-00232798
- PF-00232798 400 mg (Active Comparator)
  Interventions: Drug: PF-00232798
- PF-00232798 5 mg (Active Comparator)
  Interventions: Drug: PF-00232798
- PF-00232798 20 mg (Active Comparator)
  Interventions: Drug: PF-00232798
- PF-00232798 150 mg (Active Comparator)
  Interventions: Drug: PF-00232798

INTERVENTIONS:
Drug: PF-00232798 — Solution, 20 mg. once daily, 10 days
  Arms: PF-00232798 20 mg
Drug: PF-00232798 — Solution, 150 mg. once daily, 10 days
  Arms: PF-00232798 150 mg
Drug: PF-00232798 — Solution, 5 mg. once daily, 10 days
  Arms: PF-00232798 5 mg
Drug: PF-00232798 — Solution, 40 mg. once daily, 10 days
  Arms: PF-00232798 40 mg
Drug: PF-00232798 — Solution, 300 mg. once daily, 10 days
  Arms: PF-00232798 300 mg
Drug: PF-00232798 — Solution, 400 mg. once daily, 10 days
  Arms: PF-00232798 400 mg

SUMMARY:
To assess the viral load response, safety, tolerability and pharmacokinetics of multiple oral doses of PF 00232798 in HIV-positive patient volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic HIV-1 infected male patients between the ages of 18 and 55 years inclusive.
* Patients with CCR5 tropic virus as determined by the Monogram PhenoSense Entry assay.

Exclusion Criteria:

* Patients who have received any experimental drug within the past four months (prior to the first dosing day of the study) or who have previously received another CCR5 antagonist.
* Patients with evidence of decompensated liver disease.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Germany (2):
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Frankfurt am Main

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7691009&StudyName=A%20Phase%202%20Study%20Of%20PF-00232798%20In%20HIV%20Positive%20Patients.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to PF-00232798 oral solution once daily up to Day 10 and were followed up to Day 25 in Stage 1.
- PF-00232798 5 mg: Participants received PF-00232798 5 milligram (mg) oral solution once daily up to Day 10 and were followed up to Day 25 in Stage 1.
- PF-00232798 20 mg: Participants received PF-00232798 20 mg oral solution once daily up to Day 10 and were followed up to Day 25 in Stage 1.
- PF-00232798 150 mg: Participants received PF-00232798 150 mg oral solution once daily up to Day 10 and were followed up to Day 25 in Stage 1.
- PF-00232798 40 mg: Participants received PF-00232798 40 mg oral solution once daily up to Day 10 and were followed up to Day 25 in Stage 2.
- PF-00232798 300 mg: Participants received PF-00232798 300 mg oral solution once daily up to Day 10 and were followed up to Day 25 in Stage 2.
- PF-00232798 400 mg: Participants received PF-00232798 400 mg oral solution once daily up to Day 10 and were followed up to Day 25 in Stage 2.
Period: Stage 1 (25 Days)
Arm/Group | Placebo | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 150 mg | PF-00232798 40 mg | PF-00232798 300 mg | PF-00232798 400 mg
Started | 2 | 6 | 6 | 6 | 0 | 0 | 0
Completed | 2 | 6 | 5 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Stage 2 (25 Days)
Arm/Group | Placebo | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 150 mg | PF-00232798 40 mg | PF-00232798 300 mg | PF-00232798 400 mg
Started | 0 | 0 | 0 | 0 | 8 | 8 | 7
Completed | 0 | 0 | 0 | 0 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-00232798 400mg: Participants received PF-00232798 400 mg oral solution once daily up to Day 10 and were followed up to Day 25 in Stage 2.
- Total: Total of all reporting groups
Arm/Group | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 40 mg | PF-00232798 150 mg | PF-00232798 300 mg | PF-00232798 400mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 8 | 7 | 2 | 43
Age Continuous [Mean (Standard Deviation); unit: years] | 31.5 (8.9) | 39.8 (8.5) | 36.5 (5.4) | 36.2 (9.1) | 36.1 (9.6) | 32.9 (5) | 29 (5.7) | 35.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 8 | 6 | 8 | 7 | 2 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log 10-transformed Human Immunodeficiency Virus (HIV) Viral Load at Day 11
Description: Viral load was determined using the Roche COBAS Taqman HIV-1 assay with a lower limit of detection of 40 copies per milliliter (copies/mL). Samples with an initial reading of less than 1,000,000 copies/mL were diluted into range and re-assayed.
Time Frame: Baseline, Day 11
Population: Pharmacodynamic population included all participants who were randomized, treated and had at least 1 post-dose HIV viral load measurement in the study.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 40 mg | PF-00232798 150 mg | PF-00232798 300 mg | PF-00232798 400 mg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 6 | 8 | 7 | 2
log10 copies/mL
  Baseline | 4.692 (0.3075) | 4.338 (0.4753) | 4.306 (0.8241) | 4.483 (0.4322) | 4.315 (0.6120) | 4.715 (0.3153) | 4.482 (0.9800)
  Change at Day 11 | -0.253 (0.3308) | -0.687 (0.4260) | -0.916 (0.4267) | -1.325 (0.3887) | -1.546 (0.3028) | -1.492 (0.5103) | -0.135 (0.0089)

2. Secondary Outcome: Number of Participants With Time to Rebound of Human Immunodeficiency Virus (HIV) Viral Load
Description: The time to rebound of viral load was calculated as the time from the last dose to the time of the first occasion at which the viral load was greater than the baseline value. Results are reported for number of participants who rebound within specified days from last dose and who did not rebound up to Day 25.
Time Frame: Day 1 up to Day 25
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 40 mg | PF-00232798 150 mg | PF-00232798 300 mg | PF-00232798 400 mg | Placebo
Number analyzed (Participants) | 6 | 5 | 8 | 6 | 8 | 7 | 2
participants
  Rebound within 2 days | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Rebound within 3 days | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Rebound within 5 days | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Rebound within 9 days | 0 | 1 | 2 | 1 | 1 | 0 | 0
  Rebound within 12 days | 0 | 2 | 0 | 0 | 0 | 1 | 0
  Rebound within 15 days | 0 | 1 | 0 | 1 | 1 | 0 | 0
  No Rebound | 1 | 1 | 6 | 4 | 6 | 6 | 1

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 hour (pre-dose) on Day 1 to 9; 0 hour (pre-dose), 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 10; Day 12, 13, 15 morning
Population: Pharmacokinetic parameter analysis population included all participants who were randomized, treated and had at least 1 of the pharmacokinetic parameters of interest in the study.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 40 mg | PF-00232798 150 mg | PF-00232798 300 mg | PF-00232798 400 mg
Number analyzed (Participants) | 6 | 5 | 8 | 6 | 8 | 7
nanogram per milliliter (ng/mL) | 25.21 (13.964) | 185.57 (268.401) | 379.27 (239.376) | 2675.57 (860.860) | 3793.01 (285.845) | 4802.57 (2025.429)

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 40 mg | PF-00232798 150 mg | PF-00232798 300 mg | PF-00232798 400 mg
Number analyzed (Participants) | 6 | 5 | 8 | 6 | 8 | 7
hours | 3.0000 [1.000 to 6.000] | 1.0330 [1.000 to 3.000] | 4.0000 [1.000 to 4.000] | 3.0415 [2.000 to 4.000] | 2.0000 [2.000 to 4.000] | 2.0000 [1.000 to 3.000]

5. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Description: AUCtau= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to the time end of dosing interval (24 hours post-dose).
Time Frame: 0 hour (pre-dose), 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 10
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 40 mg | PF-00232798 150 mg | PF-00232798 300 mg | PF-00232798 400 mg
Number analyzed (Participants) | 6 | 5 | 8 | 6 | 8 | 7
nanogram*hour per milliliter (ng*hr/mL) | 265.3 (181.46) | 1157.4 (884.12) | 2945.1 (1548.47) | 17319.1 (7529.14) | 28347.9 (5435.54) | 41027.3 (20326.95)

6. Other Pre Specified Outcome: Number of Participants With Viral Tropism and Resistance
Description: Virus tropism was determined using the Monogram PhenoSense Entry assay; standard Trofile tropisim assay was used for Stage 1 and enhanced sensitivity Trofile tropisim assay was used for Stage 2.
Time Frame: Screening, pre-dose on Day 1; Day 11, 25
Population: Results for this outcome was not reported because data was collected in individual participant listings, but not summarized for analyses.
Arm/Group | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 40 mg | PF-00232798 150 mg | PF-00232798 300 mg | PF-00232798 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Chemokine Receptor 5 (CCR5) Delta 32 Genotyping and Immunophenotyping
Description: CCR5 Delta 32 genotyping and immunophenotyping was to be done to assess CCR5 Delta 32 status, other CCR5 polymorphisms, enzymes involved in drug metabolism and/or drug transport proteins in order to measure the impact of genetic variation with respect to PF-00232798 in case any unusual patterns of response or an unexplained excess of adverse events occurred.
Time Frame: Pre-dose on Day 1
Population: Results for this outcome were not analyzed because there were no unusual patterns of response or an unexplained excess of adverse events that warranted genotyping.
Arm/Group | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 40 mg | PF-00232798 150 mg | PF-00232798 300 mg | PF-00232798 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-00232798 5 mg | PF-00232798 20 mg | PF-00232798 40 mg | PF-00232798 150 mg | PF-00232798 300 mg | PF-00232798 400mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/8 | 0/6 | 0/8 | 1/7 | 0/2
Other Adverse Events (participants affected / at risk) | 2/6 | 6/6 | 7/8 | 5/6 | 6/8 | 3/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00232798 5 mg (N=6) | PF-00232798 20 mg (N=6) | PF-00232798 40 mg (N=8) | PF-00232798 150 mg (N=6) | PF-00232798 300 mg (N=8) | PF-00232798 400mg (N=7) | Placebo (N=2)
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angiopathy (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00232798 5 mg (N=6) | PF-00232798 20 mg (N=6) | PF-00232798 40 mg (N=8) | PF-00232798 150 mg (N=6) | PF-00232798 300 mg (N=8) | PF-00232798 400mg (N=7) | Placebo (N=2)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Panophthalmitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 0 | 4 | 0 | 0
Hunger (General disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 3 | 2 | 0 | 2 | 1
Hypersomnia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.